CLINICAL TRIAL: NCT06482476
Title: Medical Students' Evaluation of Dyslipidemia and LIPoprotein(a) Study (MEDLIP Study)
Brief Title: Medical Students' Evaluation of Dyslipidemia and LIPoprotein(a) Study
Acronym: MEDLIP
Status: Recruiting | Type: Observational
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Fotios Barkas, Fotios Barkas, MD, MSc, PhD, Assistant Professor of Internal Medicine Faculty of Medicine, School of Health Sciences, University of Ioannina, Ioannina, Greece, University of Ioannina
Other Study IDs: MEDLIP Study
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Insight Into the Prevalence of Elevated Lp(a) Among Greek Medical Students

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Med students: Medical students in whom Lp(a) levels will be measured
  Interventions: Diagnostic Test: Measurement of Lp(a) levels

INTERVENTIONS:
Diagnostic Test: Measurement of Lp(a) levels — Collection of a venous blood sample for the measurement of Lp(a) levels using standardized laboratory methods

SUMMARY:
This cross-sectional study aims to determine the prevalence of elevated Lp(a) levels among volunteer medical students at the Faculty of Medicine, University Hospital of Ioannina, Greece. Data collected will include demographic information, family and medical history, as well as lifestyle habits, and the study aims to provide valuable insights into the prevalence of elevated Lp(a) among Greek medical students.

DETAILED DESCRIPTION:
Lipoprotein(a) [Lp(a)] has emerged as a prevalent monogenetic cardiovascular risk factor globally. Despite its significance, clinical attention for elevated Lp(a) is suboptimal. This cross-sectional study aims to determine the prevalence of elevated Lp(a) levels among volunteer medical students at the Faculty of Medicine, University Hospital of Ioannina, Greece, as well as gather data on the demographic characteristics and medical history of this population. Statistical analysis will assess Lp(a) levels, prevalence, and associations with demographic and cardiovascular risk factors. The study aims to provide valuable insights into the prevalence of elevated Lp(a) among Greek medical students, emphasizing the importance of awareness, early diagnosis, and management of this cardiovascular risk factor.

ELIGIBILITY:
Inclusion Criteria:

* Medical students at the Faculty of Medicine, University Hospital of Ioannina, Greece.

Exclusion Criteria:

* Inability/unwillingness to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteer medical students at the Faculty of Medicine, University Hospital of Ioannina, Greece
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Lp(a) elevated | At time of measurement
Lp(a) beneath cut-off | At time of measurement

CONTACTS AND LOCATIONS:
Overall Officials: Fotios Barkas, MD, PhD, Principal Investigator — University of Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: Undecided